CLINICAL TRIAL: NCT02265276
Title: A Prospective, Randomized Trial to Compare saroGLitazar With pioglitAZone in Nonalcoholic Fatty livEr Disease (GLAZED Trial)
Brief Title: A Prospective, Randomized Trial to Compare saroGLitazar With pioglitAZone in Nonalcoholic Fatty livEr Disease
Acronym: GLAZED
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Command Hospital, India (Other Government)
Responsible Party: Principal Investigator, Hari Kumar, Endocrinologist, Command Hospital, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENDO/2014/4
Record Dates: First submitted 2014-10-07; First posted 2014-10-15 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Fatty Liver
Keywords: NAFLD, Diabetes, Glitazone
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease; Diabetes Mellitus | interventions — saroglitazar; Pioglitazone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saroglitazar Group (Active Comparator): Tab Saroglitazar 4 mg oral daily fixed dose for 24 weeks
  Interventions: Drug: Saroglitazar
- Pioglitazone Group (Placebo Comparator): Tab Pioglitazone 30 mg daily fixed dose for 24 weeks
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Saroglitazar — Tab Saroglitazar 4 mg oral daily for 24 weeks
  Other Names: Glitazar group
  Arms: Saroglitazar Group
Drug: Pioglitazone — Tab Pioglitazone 30 mg oral daily for 24 weeks
  Other Names: Placebo Comparator group
  Arms: Pioglitazone Group

SUMMARY:
Non Alcoholic Fatty Liver Disease (NAFLD) is considered as the component of metabolic syndrome. The prevalence of the same has been increasing rapidly in India, along with an increase in the prevalence of diabetes and obesity. Insulin resistance is the key underlying pathogenetic mechanism of NAFLD. NAFLD accounts for significant morbidity and mortality and the therapeutic options are limited. Insulin sensitizing drugs are used in the management of NAFLD.

DETAILED DESCRIPTION:
The therapeutic options for the management of nonalcoholic fatty liver disease (NAFLD) include lifestyle modifications, insulin sensitizers, vitamin E, antioxidants and cytoprotective agents. Glitazones are insulin sensitizing drugs and act by stimulating the PPAR gamma receptors. The drugs like Pioglitazone and Rosiglitazone have shown conflicting results in the NAFLD trials. Dual PPAR stimulators (PPAR gamma and PPAR alfa) are known as the "Glitazars" and are useful in simultaneously controlling the hyperglycemia, dyslipidemia and insulin resistance. Saroglitazar is the first drug approved in the investigators country for the management of diabetic dyslipidemia. The investigators plan to study the efficacy of this drug in comparison to Pioglitazone in patients of NAFLD over a period of 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Drug naive patients with NAFLD diagnosed on ultrasonography, BMI > 23 kg/m2 and ALT > 1.5 times the upper limit of normal

Exclusion Criteria:

* Use of any drugs other than lifestyle modification for NAFLD, HbA1c > 8% FBS>200, Bilirubin > 1.5 mg/dL
* Any illness likely to cause transaminitis and positive viral markers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Change in the NAFLD fibrosis score | At baseline and the end of 24 weeks

SECONDARY OUTCOMES:
Change in body composition | At baseline and the end of 24 weeks
Change in insulin resistance | At baseline and the end of 24 weeks
Change in lipid profile | At baseline and the end of 24 weeks
Change in HbA1c | At baseline and the end of 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hari Kumar, MD, Principal Investigator — Command Hospital
Locations (1):
- Command Hospital, Panchkula, Haryana, India